CLINICAL TRIAL: NCT02318940
Title: Comparison of Effectiveness and Safety of Two Methods for Installing Femoral Central Venous Catheters in Pediatric Intensive Care Units : Anatomical Method vs Ultrasound in Real Time.
Brief Title: Femoral Central Venous Access Comparison of 2 Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Pietro Pietroboni Fuster, Medico Pediatra, University of Chile
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRR001
Record Dates: First submitted 2014-12-12; First posted 2014-12-17 (Estimated); Results first posted 2016-12-15 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-02

CONDITIONS: Child
Keywords: ultrasound guided; femoral vein; central venous catheter; pediatric
MeSH Terms: interventions — Central Venous Catheters

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Landmark method (Other): installation of Central venous catheter In this arm the catheter will be installed under the usual method guided by anatomical landmarks.
  access will be through the femoral vein only
  Interventions: Device: central venous catheter
- Ultrasound method (Active Comparator): installation of Central venous catheter This arm of the catheter is installed using real-time ultrasound. Access will be through the femoral vein only
  Interventions: Device: central venous catheter

INTERVENTIONS:
Device: central venous catheter — installation of Central venous catheter ultrasound guided
  Arms: Ultrasound method
Device: central venous catheter — installation of Central venous catheter landmark guided
  Arms: Landmark method

SUMMARY:
The purpose of this study is to compare the effectiveness and safety of the installation of femoral central venous catheter (CVC) ultrasound-guided real-time 2D versus the landmark method

DETAILED DESCRIPTION:
STUDY DESIGN Multicenter prospective randomized study in pediatric intensive care units of the Roberto del Rio's hospital and Exequiel González Cortés' hospital. Patients from entering the study between the months of January/2015 to December/2015, after signing informed by their parents or legal guardian consent, this will be implemented by the resident

PATIENTS Previous studies report an average success rate of 50% on the first attempt in the anatomical method, both children and adults. Sample size is determined to improve on a 30% success rate using the ultrasound method. For a power of 80% in relation to success at the first attempt and with a confidence level of 95%, a total of 50 patients per branch is determined.

Method of randomization Using computer program the patient leaving 50 patients in the group with the anatomical method, and 50 patients in the ultrasound method are randomized .

OPERATOR Both installation landmark and ultrasound guidance will be performed by 3 or 4 team doctors resident in each center , who count on ≥ 3 years of experience in ICU and training in ultrasound-guided access .

DEFINITIONS

* Successful cannulation: is considered successful installation when the guide is installed without difficulty in femoral vein.
* Cannulation the first try: is considered successful when installing the CVC is accomplished by first transcutaneous passage to the glass needle .
* Attempt to cannulation: considered attempt the passage of the needle without removing or redirect moving forward. Each successive removal or redirection with a forward motion is considered more a try.
* Arterial puncture: Arterial puncture aspiration involves pulsatile arterial blood .
* Rescue: After the fifth attempt in the landmark method will change the method under ultrasound guidance and is considered not successful cannulation. Result of not having puncture site is changed.

INSTALLATION METHOD

* Anatomical : In supine with external rotation and abduction of the lower extremity is located by palpating the femoral artery in the femoral triangle and punctured medial to this towards the navel to have reflux of venous blood.
* Guided by ultrasound: Ultrasound is performed to verify the presence and proper position of a target vessel before puncturing the skin followed by real-time ultrasound to guide the needle tip during the lancing process.

OUTCOME It was considered as primary outcome main installation on the first try , and secondary outcome cannulation success, number of attempts and , as a complication of the procedure, arterial puncture. Rescue will be used after the 5th attempt in the anatomical method that will change the method under ultrasound guidance . Failure to gain access shall be considered as successful cannulation and change of puncture site

STATISTICAL ANALYSIS For statistical analysis the Stata 12.0 software was used. Continuous variables were analyzed using descriptive analysis of normal distribution with means and standard deviations , and continuous variables were not normally distributed and qualitative medians and percentiles. For the primary outcome will be used to varying dicomtómic Chi square method

ELIGIBILITY:
Inclusion Criteria:

* Need for central venous access

Exclusion Criteria:

* More than 15 years.
* Local infection at the puncture site
* Anatomical and / or functional vascular alteration known

Ages: 1 Week to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 99 (Actual)
Dates: Start 2014-12; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pietro F Pietroboni, MD, Principal Investigator — University of Chile; Cristian Carvajal, MD, Mg, Study Director — Hospital Roberto del Río
Locations (2):
- Chile (2):
  - Hospital Exequiel González Cortés, Santiago, Santiago Metropolitan
  - Hospital Roberto del Rio, Santiago, Santiago Metropolitan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu SY, Ling Q, Cao LH, Wang J, Xu MX, Zeng WA. Real-time two-dimensional ultrasound guidance for central venous cannulation: a meta-analysis. Anesthesiology. 2013 Feb;118(2):361-75. doi: 10.1097/ALN.0b013e31827bd172. PMID 23249991
- [Background] National Institute for Clinical Excellence. Guidance on the use of ultrasound locating devices for placing central venous catheters. Technology Appraisal Guidance-No.49, 2002:1-21
- [Background] American Society of Anesthesiologists Task Force on Central Venous Access; Rupp SM, Apfelbaum JL, Blitt C, Caplan RA, Connis RT, Domino KB, Fleisher LA, Grant S, Mark JB, Morray JP, Nickinovich DG, Tung A. Practice guidelines for central venous access: a report by the American Society of Anesthesiologists Task Force on Central Venous Access. Anesthesiology. 2012 Mar;116(3):539-73. doi: 10.1097/ALN.0b013e31823c9569. No abstract available. PMID 22307320
- [Background] Johnson EM, Saltzman DA, Suh G, Dahms RA, Leonard AS. Complications and risks of central venous catheter placement in children. Surgery. 1998 Nov;124(5):911-6. PMID 9823406
- [Background] Karapinar B, Cura A. Complications of central venous catheterization in critically ill children. Pediatr Int. 2007 Oct;49(5):593-9. doi: 10.1111/j.1442-200X.2007.02407.x. PMID 17875082
- [Background] Casado-Flores J, Barja J, Martino R, Serrano A, Valdivielso A. Complications of central venous catheterization in critically ill children. Pediatr Crit Care Med. 2001 Jan;2(1):57-62. doi: 10.1097/00130478-200101000-00012. PMID 12797890
- [Background] Hilty WM, Hudson PA, Levitt MA, Hall JB. Real-time ultrasound-guided femoral vein catheterization during cardiopulmonary resuscitation. Ann Emerg Med. 1997 Mar;29(3):331-6; discussion 337. doi: 10.1016/s0196-0644(97)70344-5. PMID 9055771
- [Background] Verghese ST, McGill WA, Patel RI, Sell JE, Midgley FM, Ruttimann UE. Ultrasound-guided internal jugular venous cannulation in infants: a prospective comparison with the traditional palpation method. Anesthesiology. 1999 Jul;91(1):71-7. doi: 10.1097/00000542-199907000-00013. PMID 10422930
- [Background] Verghese ST, McGill WA, Patel RI, Sell JE, Midgley FM, Ruttimann UE. Comparison of three techniques for internal jugular vein cannulation in infants. Paediatr Anaesth. 2000;10(5):505-11. doi: 10.1046/j.1460-9592.2000.00554.x. PMID 11012954
- [Background] Grebenik CR, Boyce A, Sinclair ME, Evans RD, Mason DG, Martin B. NICE guidelines for central venous catheterization in children. Is the evidence base sufficient? Br J Anaesth. 2004 Jun;92(6):827-30. doi: 10.1093/bja/aeh134. Epub 2004 Apr 30. PMID 15121722
- [Background] Karakitsos D, Labropoulos N, De Groot E, Patrianakos AP, Kouraklis G, Poularas J, Samonis G, Tsoutsos DA, Konstadoulakis MM, Karabinis A. Real-time ultrasound-guided catheterisation of the internal jugular vein: a prospective comparison with the landmark technique in critical care patients. Crit Care. 2006;10(6):R162. doi: 10.1186/cc5101. PMID 17112371
- [Background] Turker G, Kaya FN, Gurbet A, Aksu H, Erdogan C, Atlas A. Internal jugular vein cannulation: an ultrasound-guided technique versus a landmark-guided technique. Clinics (Sao Paulo). 2009;64(10):989-92. doi: 10.1590/S1807-59322009001000009. PMID 19841706
- [Background] Mitre CI, Golea A, Acalovschi I, Mocan T, Caea AM, Ruta C, Mariana M. Ultrasound-guided external jugular vein cannulation for central venous access by inexperienced trainees. Eur J Anaesthesiol. 2010 Mar;27(3):300-3. doi: 10.1097/EJA.0b013e328333c2d6. PMID 19935072
- [Background] Prabhu MV, Juneja D, Gopal PB, Sathyanarayanan M, Subhramanyam S, Gandhe S, Nayak KS. Ultrasound-guided femoral dialysis access placement: a single-center randomized trial. Clin J Am Soc Nephrol. 2010 Feb;5(2):235-9. doi: 10.2215/CJN.04920709. Epub 2009 Dec 3. PMID 19965532
- [Background] Fragou M, Gravvanis A, Dimitriou V, Papalois A, Kouraklis G, Karabinis A, Saranteas T, Poularas J, Papanikolaou J, Davlouros P, Labropoulos N, Karakitsos D. Real-time ultrasound-guided subclavian vein cannulation versus the landmark method in critical care patients: a prospective randomized study. Crit Care Med. 2011 Jul;39(7):1607-12. doi: 10.1097/CCM.0b013e318218a1ae. PMID 21494105
- [Background] Yonei A, Nonoue T, Sari A. Real-time ultrasonic guidance for percutaneous puncture of the internal jugular vein. Anesthesiology. 1986 Jun;64(6):830-1. doi: 10.1097/00000542-198606000-00033. No abstract available. PMID 3717653
- [Background] Weiner MM, Geldard P, Mittnacht AJ. Ultrasound-guided vascular access: a comprehensive review. J Cardiothorac Vasc Anesth. 2013 Apr;27(2):345-60. doi: 10.1053/j.jvca.2012.07.007. Epub 2012 Sep 18. No abstract available. PMID 22995457
- [Background] Iwashima S, Ishikawa T, Ohzeki T. Ultrasound-guided versus landmark-guided femoral vein access in pediatric cardiac catheterization. Pediatr Cardiol. 2008 Mar;29(2):339-42. doi: 10.1007/s00246-007-9066-2. Epub 2007 Sep 13. PMID 17851631
- [Background] Aouad MT, Kanazi GE, Abdallah FW, Moukaddem FH, Turbay MJ, Obeid MY, Siddik-Sayyid SM. Femoral vein cannulation performed by residents: a comparison between ultrasound-guided and landmark technique in infants and children undergoing cardiac surgery. Anesth Analg. 2010 Sep;111(3):724-8. doi: 10.1213/ANE.0b013e3181e9c475. Epub 2010 Jul 2. PMID 20601450
- [Background] McGee DC, Gould MK. Preventing complications of central venous catheterization. N Engl J Med. 2003 Mar 20;348(12):1123-33. doi: 10.1056/NEJMra011883. No abstract available. PMID 12646670
- [Background] Mansfield PF, Hohn DC, Fornage BD, Gregurich MA, Ota DM. Complications and failures of subclavian-vein catheterization. N Engl J Med. 1994 Dec 29;331(26):1735-8. doi: 10.1056/NEJM199412293312602. PMID 7984193
- [Background] Klerk CP, Smorenburg SM, Buller HR. Thrombosis prophylaxis in patient populations with a central venous catheter: a systematic review. Arch Intern Med. 2003 Sep 8;163(16):1913-21. doi: 10.1001/archinte.163.16.1913. PMID 12963564
- [Background] Lamperti M, Bodenham AR, Pittiruti M, Blaivas M, Augoustides JG, Elbarbary M, Pirotte T, Karakitsos D, Ledonne J, Doniger S, Scoppettuolo G, Feller-Kopman D, Schummer W, Biffi R, Desruennes E, Melniker LA, Verghese ST. International evidence-based recommendations on ultrasound-guided vascular access. Intensive Care Med. 2012 Jul;38(7):1105-17. doi: 10.1007/s00134-012-2597-x. Epub 2012 May 22. PMID 22614241

RESULTS

PARTICIPANT FLOW:
Groups:
- Landmark Method: installation of Central venous catheter In this arm the catheter will be installed under the usual method guided by anatomical landmarks.
  access will be through the femoral vein only
  central venous catheter: installation of Central venous catheter landmark guided
Period: Overall Study
Arm/Group | Landmark Method | Ultrasound Method
Started | 50 (in the last patient we lost the record.) | 50
Completed | 49 | 50
Not Completed | 1 | 0
Not completed — lost the record | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Landmark Method | Ultrasound Method | Total
Number analyzed (Participants) | 49 | 50 | 99
Age, Continuous [Median (Full Range); unit: months] | 12 [1 to 180] | 14 [1 to 168] | 13 [1 to 180]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 22 | 44
  Male | 27 | 28 | 55
weight [Median (Full Range); unit: kg] | 10 [3 to 113] | 9 [3 to 70] | 10 [3 to 113]

OUTCOME MEASURES:

1. Primary Outcome: Installation on the First Try
Description: Percentage of Participants with successful installation on the first transcutaneous passage of the glass needle
Time Frame: intraoperative, an average of 1 hour
Measure: Number; unit: percentage of participants
Arm/Group | Landmark Method | Ultrasound Method
Number analyzed (Participants) | 49 | 50
percentage of participants | 18 | 42

2. Secondary Outcome: Successful Installation
Description: Percentage of participants with successful installation of guide without difficulty in the femoral vein
Time Frame: intraoperative, an average of 1 hour
Measure: Number; unit: percentage of participants
Arm/Group | Landmark Method | Ultrasound Method
Number analyzed (Participants) | 49 | 50
percentage of participants | 51 | 84

3. Secondary Outcome: Number of Attempts
Description: Number of participants who succeeded in the installation of cvc in one, two, three, four or five attempts.
Time Frame: intraoperative, an average of 1 hour
Measure: Number; unit: participants
Arm/Group | Landmark Method | Ultrasound Method
Number analyzed (Participants) | 49 | 50
participants
  first attempt | 9 | 21
  second attempt | 4 | 18
  third attempt | 6 | 4
  fourth attempt | 2 | 0
  fifth attempt | 4 | 0
  Unsuccessful cannulation | 24 | 7

4. Secondary Outcome: Arterial Puncture
Description: Percentage of participants with Arterial puncture aspiration
Time Frame: intraoperative, an average of 1 hour
Measure: Number; unit: percentage of participants
Arm/Group | Landmark Method | Ultrasound Method
Number analyzed (Participants) | 49 | 50
percentage of participants | 25 | 10

ADVERSE EVENTS:
Arm/Group | Landmark Method | Ultrasound Method
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/50
Other Adverse Events (participants affected / at risk) | 0/49 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No